CLINICAL TRIAL: NCT07200323
Title: Prevalence of Postpartum Depression Among Patients of the CHUM GARE Clinic
Acronym: PPD-GARE
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2026-13020
Record Dates: First submitted 2025-09-15; First posted 2025-10-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Post-partum Depression; Maternal Health; Mental Health Issue
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postpartum depression (PPD) is a frequent complication of the postnatal period but remains underdetected in routine clinical practice. This prospective clinical study, conducted at the high-risk pregnancy clinic of the CHUM, aims to estimate the prevalence of PPD among patients seen in postpartum follow-up. It also assesses the feasibility of implementing a standardized screening protocol that combines the administration of the Edinburgh Postnatal Depression Scale (EPDS) with a clinical decision-support algorithm to guide appropriate medical follow-up. The study also seeks to explore clinical characteristics associated with higher EPDS scores.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a common complication in the weeks following childbirth, with potential consequences for maternal health and early infant development. Although validated tools such as the Edinburgh Postnatal Depression Scale (EPDS) exist, systematic screening is not uniformly integrated into routine postpartum care. This prospective observational study aims to evaluate the implementation of a structured protocol for the identification and referral of postpartum depression in a high-risk obstetric population.

The study will include 100 postpartum patients followed at the high-risk pregnancy clinic of the CHUM. All participants will be systematically screened for symptoms of postpartum depression using the EPDS during their scheduled postpartum visit. For patients with a score of 13 or higher, medical orientation will be guided by a standardized clinical algorithm that defines the recommended follow-up. Two follow-up telephone calls will be conducted, at two weeks and six weeks after the initial screening, to confirm whether the recommended referrals have been completed and to evaluate the time required to access appropriate services.

The primary objective of the study is to estimate the prevalence of postpartum depression in this population. The secondary objective is to assess the feasibility of implementing a systematic screening protocol combined with a clinical algorithm to guide referral and follow-up. The study also seeks to explore clinical characteristics associated with elevated EPDS scores, including age, level of education, lifestyle habits (smoking, alcohol or drug consumption), psychiatric, medical and obstetric history (including history of miscarriage), mode of delivery and method of perinatal analgesia, iron-deficiency anemia or iron deficiency, obstetric, anesthetic, or neonatal complications, and skin-to-skin contact in the delivery room within the first 24 hours after birth.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more
* Gave birth in the last 2 months
* Ability to understand French or English and complete the EPDS questionnaire
* Physically present at their post-partum visit at the clinic

Exclusion Criteria:

* Inability to comprehend and/or complete the EPDS
* Declines participation or does not provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who gave birth in the last 2 months at CHUM
Study Population: Patients of the high-risk pregnancy clinic (GARE - Grossesse à risque élevé) of the Centre hospitalier de l'Université de Montréal (CHUM) coming in for their post-partum visit with obstetrician
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of postpartum depression in the study population | Baseline EPDS score (Day 0)
  Proportion of patients with an EPDS score ≥13 at the 4 to 8-week postpartum visit. The Edimburgh Postnatal Depression Scale (EPDS) is a validated 10-item questionnaire designed to identify symptoms of depression in postnatal mothers. Each question asks about feelings and experiences over the past seven days, covering various emotional and psychological aspects related to perinatal mood. For each question, there are four possible responses, scored from 0 to 3, with higher numbers indicating more severe symptoms. The total EPDS score indicates the severity of potential depressive symptoms: a score of 13 or above often suggests a high risk of developing a depressive disorder.

SECONDARY OUTCOMES:
Orientation to a medical or psychosocial resource based on EPDS score and decision algorithm | Immediately after EPDS completion
  Categorical outcome measuring the type of referral initiated following EPDS screening (e.g., pamphlet of information, primary care health services, psychiatrist, primary care physician, emergency department).
Repeat EPDS score at 2-week follow-up (for scores between 13 and 16 only) | 2 weeks after initial EPDS score
  EPDS score collected by telephone at 2 weeks for patients with a Day 0 score between 13 and 16. Outcome measured as the proportion of patients whose score remains ≥13. The Edimburgh Postnatal Depression Scale (EPDS) is a validated 10-item questionnaire designed to identify symptoms of depression in postnatal mothers.
Number of days before the first contact with referred service | Assessed at two-week and, if needed, six-week follow-up calls
  Number of days between the initial referral (Day 0) and confirmed access to the referred service (by patient report).
Clinical and obstetrical factors associated with EPDS ≥13 | Chart review conducted following Day 0 visit and consent
  Exploratory analysis to evaluate associations between an elevated EPDS score (≥13) and selected clinical variables, including age, level of education, lifestyle habits (smoking, alcohol or drug consumption), psychiatric, medical and obstetric history (including history of miscarriage), mode of delivery and method of perinatal analgesia, iron-deficiency anemia or iron deficiency, obstetric, anesthetic, or neonatal complications, and skin-to-skin contact in the delivery room within the first 24 hours after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lavoie, MD, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada